CLINICAL TRIAL: NCT04726774
Title: Hypnosis for Fear of Falling in Hospitalized Older Adults? : a Feasibility Randomized Controlled Study.
Brief Title: Hypnosis for Fear of Falling in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Andrea Trombetti, Professor Andrea Trombetti, MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BASEC 2018-01550; SNCTP000003110 (Registry Identifier: SNCTP)
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Rehabilitation; Fear of Falling; Older Adults
Keywords: hypnosis; fear of falling; rehabilitation; older adults; feasibility study
MeSH Terms: interventions — Hypnosis; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental): The intervention consisted of two hypnosis sessions by a physician trained in medical hypnosis. The hypnosis group received also the usual rehabilitation program.
  Interventions: Behavioral: Hypnosis; Behavioral: Rehabilitation program
- Control group (Active Comparator): The control group follow the usual rehabilitation program which includes intensive physiotherapy for 2 weeks (i.e., focused on walking and enhancing balance exercises in group or individual and group) and patient education on the risk of falling and on prevention of falls.
  Interventions: Behavioral: Rehabilitation program

INTERVENTIONS:
Behavioral: Hypnosis — Two sessions of hypnosis, about 30 minutes each, weekly provided, by a physician trained in medical hypnosis.
  Each session was realized as possible during walking, according to the agreement and the physical status of the participant.
  Each sessions of hypnosis includes 3 phases : induction, walk perception alteration and post-hypnotic suggestion.
  Arms: Hypnosis group
Behavioral: Rehabilitation program — Intensive physiotherapy for 2 weeks, with walking and balance exercises, (individual and group exercises). Education of risk of falling and prevention of falls.

SUMMARY:
Fear of falling is associated with numerous negative health outcomes in older adults and can limit rehabilitation. Few treatments are effective in fear of falling. Hypnosis is now recognized as an effective treatment for a variety of conditions, especially anxiety and pain, which can be integrated safely with conventional medicine. Therefore, the objective was to assess the feasibility of a randomized controlled trial to examine whether hypnosis reduces fear of falling in an inpatient geriatric population. In this randomized pilot trial, patients hospitalized in geriatric rehabilitation wards were randomly allocated to either an intervention group (hypnosis plus usual rehabilitation program) or a control group (usual rehabilitation program only). Primary feasibility outcomes were recruitment rate, retention rate, and adherence to the intervention. Secondary outcomes concerned the impact of hypnosis in rehabilitation in fear of falling scores, functional scores, length of stay, and drugs.

DETAILED DESCRIPTION:
This single-center randomized controlled feasibility trial was conducted in a 296 beds acute care and rehabilitation geriatric hospital of Geneva University Hospitals (Switzerland).

After consent, patients were randomized to either the intervention group or the control group. The randomization sequence was computer-generated (ratio 1:1) and concealed until official patient enrolment. All study staff members, including physiotherapists and occupational therapists, were blinded to group allocation, with the exception of the hypnotherapist. All statistical analyses were performed by a blinded statistician.

The intervention consisted of two hypnosis sessions of about 30 minutes, weekly provided, by a physician trained in medical hypnosis. Each session was realized as possible during walking, according to the agreement and the physical status of the participant. The intervention was provided in the complement of the usual rehabilitation program. Both the intervention and control groups received the usual rehabilitation program, a multifactorial fall-and-fracture risk-based assessment, and management intervention, which has been shown to be effective in improving physical parameters related to the risk of fall and disability among high-risk oldest-old patients. This program includes intensive physiotherapy for 2 weeks (i.e., focused on walking and enhancing balance exercises in group or individual and group) and patient education on the risk of falling and on prevention of falls.

The target sample size was 30 participants (15 participants in each group, pilot study). The study was approved by the State of Geneva's Ethics Committee (2018-01550). All patients provided written informed consent before any study-related procedure.

The feasibility of a randomized controlled trial with hypnosis in rehabilitation was assessed by recruitment rate, retention rate, adherence to hypnosis, and adverse events.

Fear of falling was assessed by different validated scales. Each scale was completed by each participant three times (week 0 (at baseline): before intervention; week 1 (during intervention): between the two hypnosis sessions; week 2 (at the end of the study): after all interventions), with or without the help of the occupational therapist.

Descriptive statistics were reported as mean ± standard deviation or number (percent). The hypnosis and the control groups were compared at baseline using t-tests or Fisher's exact test as appropriate. Longitudinal data were analyzed according to the intention-to-treat concept. Longitudinal data for fear of falling scores, Functional Independence Measure score, and Short Physical Performance Battery score, were analyzed using linear mixed-effects regression models, a negative binomial model for in-hospital falls, and t-tests for medications and length of stay. The incidence of in-hospital falls during hospital stay was analyzed using a negative binomial regression model.

ELIGIBILITY:
Inclusion Criteria:

* admitted in a rehabilitation program specialized in falls and fracture risk assessment and management
* 65 years and over

Exclusion Criteria:

* psychiatrics disorders
* did not speak french
* lacking decisional capacity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | through study completion, an average of 6 months
  recruitement rate was defined by the number of included patients dividing by the number of weeks it takes to include them.
feasibility of hypnosis | through study completion, an average of 6 months
  hypnosis adherence was defined by the number of total sessions of hypnosis

SECONDARY OUTCOMES:
Impact of hypnosis on fear of falling | through study completion, an average of 6 months
  by comparing scores of questionnaires validated to assess fear of falling between groups
Impact of hypnosis on functional | through study completion, an average of 6 months
  by comparing functional ability assessed by Functional Independency Measure score and Short Physical Performance Battery score between both groups
Impact of hypnosis on length of stay | through study completion, an average of 6 months
  length of stay was defined by the number of day of hospitalization, and was compared between both groups
Impact of hypnois on number of drugs | through study completion, an average of 6 months
  number of drugs at the end of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation and Geriatrics, Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuvelier C, Hars M, Zamorani-Bianchi MP, Herrmann FR, Wieczorkiewicz CD, Zekry D, Gold G, Trombetti A. Hypnosis to reduce fear of falling in hospitalized older adults: a feasibility randomized controlled trial. Pilot Feasibility Stud. 2023 Aug 9;9(1):139. doi: 10.1186/s40814-023-01366-3. PMID 37559112